CLINICAL TRIAL: NCT05025163
Title: Cost-effectiveness Analysis of Fluoride Foam and Fluoride Varnish in Preventing Dental Caries in the Primary Teeth of Preschool Children With High Caries Risk
Brief Title: Cost-effectiveness of Topical Fluoride in Preventing Deciduous Dental Caries in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Chronic and Noncommunicable Disease Control and Prevention, China CDC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCNCD
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries in Children
Keywords: cost effectiveness; fluoride foam; fluoride varnish; dental caries; clinical trial
MeSH Terms: conditions — Dental Caries | interventions — sodium fluoride topical preparation; Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): no intervention in the control group
- fluoride foam group (Experimental): intervention; fluoride foam application (with 1.23% fluoride foam application on teeth )
  Interventions: Drug: 1.23% fluoride foam application
- fluoride varnish group (Experimental): intervention; fluoride varnish application (with 2.26% fluoride varnish application on teeth)
  Interventions: Drug: 2.26% fluoride varnish application

INTERVENTIONS:
Drug: 1.23% fluoride foam application — topical application of fluoride foam every 6 months
  Other Names: fluoride foam
  Arms: fluoride foam group
Drug: 2.26% fluoride varnish application — topical application of fluoride varnish every 6 months
  Other Names: Duraphat (Colgate)
  Arms: fluoride varnish group

SUMMARY:
Fluoride foam and fluoride varnish are effectiveness in prevention deciduous dental caries. However, the relative clinical efficacy and cost-effectiveness of these two interventions are uncertain. This study aims to evaluate the relative clinical effectiveness and cost-effectiveness of fluoride foam and fluoride varnish in preventing dental caries in the primary teeth of preschool children with high caries risk.

DETAILED DESCRIPTION:
This 24-month randomized clinical trial aims to compare the clinical efficacy and cost-effectiveness of topical fluoride application of fluoride foam and fluoride varnish in preventing dental caries in the primary teeth of preschool children with high caries risk in Harbin,Heilongjiang Province,China.

Preschool children (3-4 years) with high caries risk will be invited to participant in this study. An invitation letter will be sent to the parents explaining the purpose and procedures of this study.Parental concent will be sought.

The children will be randomly divided into three groups: the control group-no intervention; the intervention group 1 - applications of 1.23% fluoride foam every 6 months; the intervention group 2- applications of 2.26% fluoride varnish every 6 months.

Dental clinical examination of the children will be performed at the beginning of the study,12 months and 24 months later.The dental examiners will receive unified training and consistency test of dental caries survey.Only when the Kappa value reached 0.8 can oral examiners participate in the oral examination.Dental caries condition will be recorded. Approximately 5% of children will be re-examined to determine the reliability of the results.

The status of any possible side/adverse effects will be recorded in the follow-up examinations.

The data of the study will be analysed by SPSS Statistical Analysis Software.The differences among the groups will be calculated and compared. And p<0.05 will be considered statistically significant.

ELIGIBILITY:
Kindergartens Inclusion Criteria:

* Kindergartens which are all located in Harbin, Heilongjiang Province, China;
* Kindergartens which are basically the same in terms of school scale, student source structure, economic level and sanitary conditions;
* Kindergartens with the same source of domestic water, or with the same fluoride concentration in water , and the fluoride concentration in water less than 1.0mg/L.

Children Inclusion Criteria:

* Children aged over 3-year and under 4-year at the time of the survey;
* Children in good health;
* Children with a certain degree of understanding and good compliance;
* Children whose parents sign the informed consent form.

Exclusion Criteria:

* Children who are unable to cooperate or have a strong vomiting reflex;
* Children with a history of asthma or allergies;
* Children with other contraindications specified in the product manual.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1083 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
The mean number of decayed,missing and filled teeth at baseline,12 months and 24 months | 24 months
  The mean number of decayed,missing and filled teeth in fluoride foam group,fluoride varnish group and control group at baseline,12 months and 24 months
The mean number of decayed,missing and filled teeth surfaces at baseline,12 months and 24 months | 24 months
  The mean number of decayed,missing and filled teeth surfaces in fluoride foam group,fluoride varnish group and control group at baseline,12 months and 24 months
The change of mean number of decayed,missing and filled teeth at baseline,12 months and 24 months | 24 months
  The change of mean number of decayed,missing and filled teeth in fluoride foam group,fluoride varnish group and control group at baseline,12 months and 24 months
The change of mean number of decayed,missing and filled teeth surfaces at baseline,12 months and 24 months | 24 months
  The change of mean number of decayed,missing and filled teeth surfaces in fluoride foam group,fluoride varnish group and control group at baseline,12 months and 24 months

SECONDARY OUTCOMES:
The mean cost per caries avoided after 12 months and 24 months | 24 months
  The mean cost per caries avoided in fluoride foam group and fluoride varnish group after 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiao Wang, Study Director — National Center for Chronic and Noncommunicable Disease Control and Prevention, China CDC

IPD SHARING:
Plan to Share IPD: No